CLINICAL TRIAL: NCT03826407
Title: Development of a Point of Care System for Automated Coma Prognosis - A Prospective Cohort Study
Brief Title: Development of a Point of Care System for Automated Coma Prognosis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Natural Sciences and Engineering Research Council, Canada (Other); Hamilton Health Sciences Corporation (Other); Brain Vision Solutions Inc. (Unknown); McGill University (Other)
Responsible Party: Sponsor
Other Study IDs: ComaML2018; CPG158287 (Other Grant/Funding Number: Canadian Institutes of Health Research); CHRP 523461-18 (Other Grant/Funding Number: Natural Sciences and Engineering Research Council)
Record Dates: First submitted 2019-01-18; First posted 2019-02-01 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Coma; Disorder of Consciousness; Minimally Conscious State; Vegetative State; Neuropathology
Keywords: Coma; Machine Learning; Prognosis; Electrophysiology; Event-related potentials; Electroencephalography; Mismatch Negativity; Auditory Brainstem Response; Disorders of Consciousness; EEG; ERP
MeSH Terms: conditions — Coma; Consciousness Disorders; Persistent Vegetative State

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DOC patients: Patients in coma (GCS score of 3-8) or with other disorder of consciousness, primarily Minimally Conscious State (MCS) or Unresponsive Wakefulness Syndrome (UWS; also known as vegetative state)
- Healthy Control: Matched healthy controls without current neurological diagnoses

SUMMARY:
Electroencephalogram/event-related potentials (EEG/ERP) data will be collected from 50 participants in coma or other disorder of consciousness (DOC; i.e., Unresponsive Wakefulness Syndrome [UWS] or Minimally Conscious State [MCS]), clinically diagnosed using the Glasgow Coma Scale (GCS). For coma patients, EEG recordings will be conducted for up to 24 consecutive hours at a maximum of 5 timepoints, spanning 30 days from the date of recruitment, to track participants' clinical state. For DOC patients, there will be an initial EEG recording up to 24 hours, with possible subsequent weekly recordings up to 2 hours. An additional dataset from 40 healthy controls will be collected, each spanning up to a 12-hour recording period in order to formulate a baseline. Collected data are to form the basis for automatic analysis and detection of ERP components in DOC, using a machine learning paradigm. Salient features (i.e., biomarkers) extracted from the ERPs and resting-state EEG will be identified and combined in an optimal fashion to give an accurate indicator of prognosis.

DETAILED DESCRIPTION:
The Problem: Coma is a state of unconsciousness with a variety of causes. Traditional tests for coma outcome prediction are mainly based on a set of clinical observations (e.g., pupillary constriction). Recently however, event-related potentials (ERPs; which are transient electroencephalogram [EEG] responses to auditory, visual, or tactile stimuli) have been introduced as useful predictors of a positive coma outcome (i.e., emergence). However, such tests require a skilled neurophysiologist, and such people are in short supply. Also, none of the current approaches has sufficient positive and negative predictive accuracies to provide definitive prognoses in the clinical setting.

Objective: The investigators will apply innovative machine learning methods to analyze patient EEGs (50 patients and 40 healthy controls) to develop a simple, objective, replicable, and inexpensive point of care system which can significantly improve the accuracy of coma prognosis relative to current methods. The physical requirements of the proposed system consist only of an EEG system (inexpensive in terms of medical equipment) and a conventional laptop computer.

Methodology: The investigators intend to extend the team's newest algorithms and develop machine learning tools for automatic analysis and detection of ERP components. Preliminary results by the team in this respect have been very promising. The most salient features (i.e., biomarkers) extracted from the ERP will be identified and combined in an optimal fashion to give an accurate indicator of prognosis. Features will be extracted from resting state brain networks and from network trajectories associated with the processing of ERP signals.

Significance: The proposed work will enable critical care physicians to assess coma prognosis with speed and accuracy. Thus, families and their health care team will be provided the most accurate information possible to guide discussions of goals of care and life-sustaining therapies in the context of dealing with the consequences of devastating neurological injury.

ELIGIBILITY:
Inclusion Criteria:

* Patients (≥ 18 years of age) primarily admitted to the Intensive Care Units, Neurological Step Down Unit, or Coronary Care Unit at Hamilton General Hospital who are in coma with Glasgow Coma Scale (GCS) score of 3-8, or;
* Patients (≥ 18 years of age) who have other disorders of consciousness, primarily Minimally Conscious State (MCS) or Unresponsive Wakefulness Syndrome (UWS; also known as vegetative state).

Exclusion Criteria:

* Severe liver failure (i.e., Child-Pugh Class C)
* Severe renal failure (i.e., Urea ≥ 40)
* Previous open-head injury
* Known primary and secondary central nervous system malignancy
* Known hearing impairment
* Previous intracranial pathology requiring neurosurgical interventions in the past 72 hours
* Anyone who is deemed medically unsuitable for this study by the attending intensivists

Healthy Controls:

Inclusion:

* ≥ 18 years of age
* no visual, language, learning, or hearing problems
* no history of neurological or psychiatric disorder
* not currently taking any medications that act on the central nervous system, such as antidepressants, anxiolytics, or anti-epileptics

Exclusion:

(During the COVID-19 pandemic only)

* ≥ 60 years of age
* have a weakened immune system
* have one or more of the COVID-19 high risk medical conditions, according to the government of Canada website: https://www.canada.ca/en/public-health/services/publications/diseases-conditions/people-high-risk-for-severe-illness-covid-19.html.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The Coma/DOC Group will include 50 patients from the Intensive Care Units, Neurological Step Down Unit, or Coronary Care Unit at Hamilton General Hospital (Ontario, Canada) who are in coma (GCS score =3-8), or who have other disorders of consciousness (MCS or UWS).
  The Control Group of 40 matched healthy controls will be recruited primarily from the Hamilton community (Ontario, Canada).
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-08-12 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change in multiple electrophysiological measures across specified time points during coma | up to 30 days from date of recruitment
  Event-related potentials (ERP) and resting state periods will be assessed at the specified intervals as a difference between successive timepoints. The ERP measures will include amplitude and latency values of N1, P2, MMN, P3a, P3b, and N400 to assess different levels of conscious processing and presence of signs of a conscious state predictive of subsequent emergence. Also, resting EEG measures will be obtained at regular intervals. EEG/ERP data will be recorded for up to 24 consecutive hours at a maximum of 5 timepoints spanning 30 days from the date of recruitment to track the participants' progression. The date of the initial assessment will be denoted as Day 0, and the subsequent assessments will take place ideally on Day 3, Day 10, Day 20 and Day 30, unless there is a ≥ 2 point of change in the patient's GCS score. Change in all specified measures will be assessed across the up to 24-hour recordings taken at 5 different timepoints.
Change in multiple electrophysiological measures across specified time points during MCS or UWS | up to 6 months from date of recruitment
  Event-related potentials (ERP) and resting state periods will be assessed at the specified intervals as a difference between successive timepoints. The ERP measures will include amplitude and latency values of N1, P2, MMN, P3a, P3b, and N400 to assess different levels of conscious processing and presence of signs of a conscious state predictive of subsequent emergence. Also, resting EEG measures will be obtained at regular intervals. EEG/ERP data will be recorded for an initial period of up to 24 consecutive hours, followed by up to 2-hour long recordings that may be conducted approximately once a week until the patient either regains full consciousness, is no longer within the Hamilton Health Sciences system, or until 6 months from the date of their enrollment into the study, whichever occurs first. Change in all specified measures will be assessed across the recordings taken at each timepoint.
Correlation between behavioral and electrophysiological measures after coma/DOC emergence | Within a 30-day time period post recruitment
  Patient emergence will be monitored using the Glasgow Outcome Scale (GOS). In the case of patient emergence, the full electrophysiological test procedures are recorded to correlate with traditional behavioral measures. The electrophysiological measures obtained at this timepoint (emergence) will be compared to the same measures obtained at the different time points during coma/DOC (Outcome 1/2) to detect both clinically relevant change and possible prognostic markers that may have been obtained at an earlier test point.
Sensitivity and specificity of prognostic capabilities of electrophysiological measures | Within a 30-day time period post recruitment
  Analyses will compare the electrophysiological measures as outcome predictors to traditional behaviorally-based tools.
Feasibility of procedure | up to 6 months from date of recruitment
  The team will also evaluate whether the repeated EEG sessions, lasting up to 24 hours, during the coma/DOC duration is a feasible approach to predict the emergence and outcome from coma.

SECONDARY OUTCOMES:
Correlation between individual patient factors, EEG results, and outcome for coma | up to 30 days from date of recruitment
  The study also collects demographic, medical history, injury information, and other physiological markers from the patient's health record and concurrent physiological assessment during the study period. Analyses will assess correlations between these factors and coma outcome and EEG findings.
Correlations between individual patient factors, EEG results, and outcome for DOC | up to 6 months from date of recruitment
  The study also collects demographic, medical history, injury information, and other physiological markers from the patient's health record and concurrent physiological assessment during the study period. Analyses will assess correlations between these factors and DOC outcome and EEG findings.

CONTACTS AND LOCATIONS:
Overall Officials: John F Connolly, PhD, Principal Investigator — McMaster University; Alison Fox-Robichaud, MD, Study Chair — Hamilton Health Sciences - Hamilton General site
Locations (1):
- McMaster University Hamilton Health Sciences / Hamilton General Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
To be decided

REFERENCES:
- [Background] Jones C. Glasgow coma scale. Am J Nurs. 1979 Sep;79(9):1551-3. No abstract available. PMID 258560
- [Background] Chiappa KH, Hill RA. Evaluation and prognostication in coma. Electroencephalogr Clin Neurophysiol. 1998 Feb;106(2):149-55. doi: 10.1016/s0013-4694(97)00118-1. PMID 9741776
- [Background] de Sousa LC, Colli BO, Piza MR, da Costa SS, Ferez M, Lavrador M. Auditory brainstem response: prognostic value in patients with a score of 3 on the Glasgow Coma Scale. Otol Neurotol. 2007 Apr;28(3):426-8. doi: 10.1097/MAO.0b013e3180326170. PMID 17303965
- [Background] Logi F, Fischer C, Murri L, Mauguiere F. The prognostic value of evoked responses from primary somatosensory and auditory cortex in comatose patients. Clin Neurophysiol. 2003 Sep;114(9):1615-27. doi: 10.1016/s1388-2457(03)00086-5. PMID 12948790
- [Background] Lew HL, Poole JH, Castaneda A, Salerno RM, Gray M. Prognostic value of evoked and event-related potentials in moderate to severe brain injury. J Head Trauma Rehabil. 2006 Jul-Aug;21(4):350-60. doi: 10.1097/00001199-200607000-00006. PMID 16915010
- [Background] Kane NM, Butler SR, Simpson T. Coma outcome prediction using event-related potentials: P(3) and mismatch negativity. Audiol Neurootol. 2000 May-Aug;5(3-4):186-91. doi: 10.1159/000013879. PMID 10859412
- [Background] Morlet D, Fischer C. MMN and novelty P3 in coma and other altered states of consciousness: a review. Brain Topogr. 2014 Jul;27(4):467-79. doi: 10.1007/s10548-013-0335-5. Epub 2013 Nov 27. PMID 24281786
- [Background] Fischer C, Morlet D, Bouchet P, Luaute J, Jourdan C, Salord F. Mismatch negativity and late auditory evoked potentials in comatose patients. Clin Neurophysiol. 1999 Sep;110(9):1601-10. doi: 10.1016/s1388-2457(99)00131-5. PMID 10479027
- [Background] Holeckova I, Fischer C, Giard MH, Delpuech C, Morlet D. Brain responses to a subject's own name uttered by a familiar voice. Brain Res. 2006 Apr 12;1082(1):142-52. doi: 10.1016/j.brainres.2006.01.089. PMID 16703673
- [Background] Garrido MI, Kilner JM, Stephan KE, Friston KJ. The mismatch negativity: a review of underlying mechanisms. Clin Neurophysiol. 2009 Mar;120(3):453-63. doi: 10.1016/j.clinph.2008.11.029. Epub 2009 Jan 31. PMID 19181570
- [Background] Sonnadara RR, Alain C, Trainor LJ. Occasional changes in sound location enhance middle latency evoked responses. Brain Res. 2006 Mar 3;1076(1):187-92. doi: 10.1016/j.brainres.2005.12.093. Epub 2006 Feb 17. PMID 16487494
- [Background] Duncan CC, Barry RJ, Connolly JF, Fischer C, Michie PT, Naatanen R, Polich J, Reinvang I, Van Petten C. Event-related potentials in clinical research: guidelines for eliciting, recording, and quantifying mismatch negativity, P300, and N400. Clin Neurophysiol. 2009 Nov;120(11):1883-1908. doi: 10.1016/j.clinph.2009.07.045. Epub 2009 Sep 30. PMID 19796989
- [Background] Schnakers C, Vanhaudenhuyse A, Giacino J, Ventura M, Boly M, Majerus S, Moonen G, Laureys S. Diagnostic accuracy of the vegetative and minimally conscious state: clinical consensus versus standardized neurobehavioral assessment. BMC Neurol. 2009 Jul 21;9:35. doi: 10.1186/1471-2377-9-35. PMID 19622138
- [Background] Guldenmund P, Stender J, Heine L, Laureys S. Mindsight: diagnostics in disorders of consciousness. Crit Care Res Pract. 2012;2012:624724. doi: 10.1155/2012/624724. Epub 2012 Nov 14. PMID 23213492
- [Background] Giacino JT, Fins JJ, Laureys S, Schiff ND. Disorders of consciousness after acquired brain injury: the state of the science. Nat Rev Neurol. 2014 Feb;10(2):99-114. doi: 10.1038/nrneurol.2013.279. Epub 2014 Jan 28. PMID 24468878
- [Background] Laureys S, Celesia GG, Cohadon F, Lavrijsen J, Leon-Carrion J, Sannita WG, Sazbon L, Schmutzhard E, von Wild KR, Zeman A, Dolce G; European Task Force on Disorders of Consciousness. Unresponsive wakefulness syndrome: a new name for the vegetative state or apallic syndrome. BMC Med. 2010 Nov 1;8:68. doi: 10.1186/1741-7015-8-68. PMID 21040571
- [Background] Armanfard N, Komeili M, Reilly JP, Mah R, Connolly JF. Automatic and continuous assessment of ERPs for mismatch negativity detection. Annu Int Conf IEEE Eng Med Biol Soc. 2016 Aug;2016:969-972. doi: 10.1109/EMBC.2016.7590863. PMID 28268485
- [Background] Ghosh-Dastidar S, Adeli H, Dadmehr N. Principal component analysis-enhanced cosine radial basis function neural network for robust epilepsy and seizure detection. IEEE Trans Biomed Eng. 2008 Feb;55(2 Pt 1):512-8. doi: 10.1109/TBME.2007.905490. PMID 18269986
- [Background] Guler I, Ubeyli ED. Multiclass support vector machines for EEG-signals classification. IEEE Trans Inf Technol Biomed. 2007 Mar;11(2):117-26. doi: 10.1109/titb.2006.879600. PMID 17390982
- [Background] Cao C, Tutwiler RL, Slobounov S. Automatic classification of athletes with residual functional deficits following concussion by means of EEG signal using support vector machine. IEEE Trans Neural Syst Rehabil Eng. 2008 Aug;16(4):327-35. doi: 10.1109/TNSRE.2008.918422. PMID 18701381
- [Background] Ravan M, Hasey G, Reilly JP, MacCrimmon D, Khodayari-Rostamabad A. A machine learning approach using auditory odd-ball responses to investigate the effect of Clozapine therapy. Clin Neurophysiol. 2015 Apr;126(4):721-30. doi: 10.1016/j.clinph.2014.07.017. Epub 2014 Aug 27. PMID 25213349
- [Background] Khodayari-Rostamabad A, Reilly JP, Hasey GM, de Bruin H, Maccrimmon DJ. A machine learning approach using EEG data to predict response to SSRI treatment for major depressive disorder. Clin Neurophysiol. 2013 Oct;124(10):1975-85. doi: 10.1016/j.clinph.2013.04.010. Epub 2013 May 15. PMID 23684127
- [Background] Wijdicks EF, Bamlet WR, Maramattom BV, Manno EM, McClelland RL. Validation of a new coma scale: The FOUR score. Ann Neurol. 2005 Oct;58(4):585-93. doi: 10.1002/ana.20611. PMID 16178024
- [Background] Jennett B, Bond M. Assessment of outcome after severe brain damage. Lancet. 1975 Mar 1;1(7905):480-4. doi: 10.1016/s0140-6736(75)92830-5. PMID 46957
- [Background] Armanfard N, Reilly JP, Komeili M. Local Feature Selection for Data Classification. IEEE Trans Pattern Anal Mach Intell. 2016 Jun;38(6):1217-27. doi: 10.1109/TPAMI.2015.2478471. Epub 2015 Sep 14. PMID 26390448
- [Background] Armanfard N, Reilly JP, Komeili M. Logistic Localized Modeling of the Sample Space for Feature Selection and Classification. IEEE Trans Neural Netw Learn Syst. 2018 May;29(5):1396-1413. doi: 10.1109/TNNLS.2017.2676101. Epub 2017 Mar 21. PMID 28333643
- [Derived] Connolly JF, Reilly JP, Fox-Robichaud A, Britz P, Blain-Moraes S, Sonnadara R, Hamielec C, Herrera-Diaz A, Boshra R. Development of a point of care system for automated coma prognosis: a prospective cohort study protocol. BMJ Open. 2019 Jul 17;9(7):e029621. doi: 10.1136/bmjopen-2019-029621. PMID 31320356